CLINICAL TRIAL: NCT03492099
Title: Assessing the Safety of Buprenorphine in People With Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00159636
Record Dates: First submitted 2018-03-27; First posted 2018-04-10 (Actual); Results first posted 2020-10-01 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Buprenorphine Arm (Experimental): This is the main and only arm of the study. All patients in this arm will undergo the steps outlined in the protocol to convert to buprenorphine treatment.
  Interventions: Drug: buprenorphine

INTERVENTIONS:
Drug: buprenorphine — Patients in this study will receive dosages to be determined by a physician that are specific to each patient.
  Other Names: Zubsolv; Suboxone; Buprenorphine Sublingual (SL)

SUMMARY:
This study will assess the safety of changing pain medications (opioids) adult sickle cell patients take to another type of medication therapy (buprenorphine). Patients will be asked questions about their quality of life. Other tools for assessment will also be administered.

DETAILED DESCRIPTION:
This is a descriptive, pilot study to assess the safety of converting a subset of adult sickle cell patients who are on effective disease modifying therapy (on high dose oral opioids who are unable to wean off opioids) and who continue to have frequent acute visits where parenteral opioids are administered to convert all opioid treatments to buprenorphine. Quality of life will be assessed using the Adult Sickle Cell Quality of life Measurement tool (ASCQ-Me), the Brief Pain Inventory (BPI), two Patient-Reported Outcomes Measurement Information System (PROMIS) surveys (short-form Pain Interference and Physical Function), and frequency of acute pain visits.

Buprenorphine is a partial mu-agonist and kappa antagonist and has a high affinity for the mu receptors with an elimination half-life of 28-37 hours for the sublingual administration. The lower risk for misuse, diminished withdrawal symptoms and cravings for opioids as well as the reduced risk of overdose make it an appealing alternative. Recent data on successful conversion for patients with chronic pain show a decrease in pain scores and increase in quality of life measurements after the beginning buprenorphine therapy for more than two months.

The first dose will be determined for each patient by a physician to ensure that the dosage of buprenorphine will be appropriate given the patient's current opioid dosage. There is the risk of withdrawal induced vaso-occlusive crisis (VOC).

Within 30 days prior to conversion to buprenorphine, a patient will take the ASCQ-Me, BPI, and two PROMIS surveys. Twenty-four hours prior to conversion, the patient will stop all opioid intake. The day of conversion, the patient will take a Clinical Opiate Withdrawal Scale (COWS) survey to determine whether they are in withdrawal. If so, the patient will begin buprenorphine conversion. They will also retake the aforementioned quality of life surveys. The patient will return on days 1, 14, 30, 90, and 180 to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Sickle Cell Disease, any genotype
* On disease modifying therapy (either chronic transfusions or hydroxyurea)
* On chronic daily full agonist opioid therapy with doses ranging from 90 to 400 morphine equivalents
* Have greater than 5 acute care visits in the last 6 months or have daily pain of 7 or higher on the Visual Analog Scale despite chronic opioid therapy.
* Able to provide consent
* Has medical insurance

Exclusion Criteria:

* Acute vaso-occlusive crisis on day of or day prior to buprenorphine initiation
* Use of methadone as long acting opioid (due to prolonged half-life and limited data in other populations)
* Use of illicit drugs as documented by urine toxicology screen (except for THC)
* Pregnancy
* Acute or severe bronchial asthma
* Hypersensitivity to buprenorphine or any component of the product
* Medical disorder, condition, or history that in the investigator's judgement would impair the patient's ability to participate or complete this study or render the patient to be inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lanzkron, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data will be published at some point in the future but individual data will not be disclosed

REFERENCES:
- [Background] Daitch D, Daitch J, Novinson D, Frey M, Mitnick C, Pergolizzi J Jr. Conversion from high-dose full-opioid agonists to sublingual buprenorphine reduces pain scores and improves quality of life for chronic pain patients. Pain Med. 2014 Dec;15(12):2087-94. doi: 10.1111/pme.12520. Epub 2014 Sep 12. PMID 25220043
- [Background] Carroll CP, Lanzkron S, Haywood C Jr, Kiley K, Pejsa M, Moscou-Jackson G, Haythornthwaite JA, Campbell CM. Chronic Opioid Therapy and Central Sensitization in Sickle Cell Disease. Am J Prev Med. 2016 Jul;51(1 Suppl 1):S69-77. doi: 10.1016/j.amepre.2016.02.012. PMID 27320469
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Wesson DR, Ling W. The Clinical Opiate Withdrawal Scale (COWS). J Psychoactive Drugs. 2003 Apr-Jun;35(2):253-9. doi: 10.1080/02791072.2003.10400007. PMID 12924748

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine Arm: This is the main and only arm of the study. This was an observational trial in which patients who were converted to buprenorphine had data collected on hospital utilization before and after conversion to buprenorphine and filled out surveys listed in secondary outcomes.
  buprenorphine: As this was part of clinical care individual dosages were dependent on prior opioid exposure and patient characteristics.
Period: Overall Study
Arm/Group | Buprenorphine Arm
Started | 47
Completed | 43
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Buprenorphine Arm
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 46
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Require Hospitalization Within 72 Hours Post Conversion From Full Agonist Opioids to Buprenorphine-based Pain Treatment
Description: Data will be collected on need for hospitalization within 72 hours of conversion due to withdrawal induced vaso-occlusive crisis (VOC). If 2 out of the first 5 patients require hospitalization within 72 hours of conversion the study will be stopped and we will assess what changes need to be made in the protocol to decrease the risk of hospitalization triggered by the conversion.
Time Frame: 72 hours after buprenorphine initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Arm
Number analyzed (Participants) | 43
Participants | 1

2. Secondary Outcome: Change in the Number of Acute Care Visits Per Subject in the 6 Months Prior to Buprenorphine (BUP) Induction and in the 6 Months Post to BUP Induction
Description: Change in the number of acute care visits per subject in the 6 months prior to BUP induction and in the 6 months post to BUP induction will be observed by comparing the mean number of acute care visits per patient- either to Emergency Department (ED) or to Sickle Cell Infusion Center - in the six months prior to BUP induction and in the six months post to BUP induction.
Time Frame: 6 months pre BUP induction, 6 months post BUP induction
Measure: Mean (Standard Deviation); unit: acute care visits per patient
Arm/Group | Buprenorphine Arm
Number analyzed (Participants) | 43
acute care visits per patient
  Number of Acute Visits per patient 6 months prior to BUP induction | 11.86 (11.92)
  Number of Acute Visits per patient 6 months post BUP induction | 3.35 (3.79)

3. Secondary Outcome: Change in Severity of Opiate Withdrawal, Based on the Clinical Opiate Withdrawal Scale (COWS) Score
Description: Change in severity of opiate withdrawal will be observed by comparing the mean COWS score at BUP induction and 1 day post induction. All patients will be in opiate withdrawal at the time of buprenorphine induction and at the end of the first day of induction. The level of withdrawal will be measured by the COWS score, an 11-item scale designed to be administered by a clinician. The score ranges from 0-4 (no withdrawal), 5-12 (mild withdrawal), 13-24 (moderate withdrawal), 25-36 (severe withdrawal), and 36-48 (most severe withdrawal).
Time Frame: COWS score at BUP induction, COWS score at the end of the first day of induction
Population: 38 out of 43 patients had complete pre-induction COWS data 37 out of 43 patients had complete post-induction COWS data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buprenorphine Arm
Number analyzed (Participants) | 38
score on a scale
  COWS score at BUP induction | 8.92 (3.8)
  COWS score at the end of the first day of induction: number analyzed (Participants) | 37
  COWS score at the end of the first day of induction | 3.32 (2.46)

4. Secondary Outcome: Number of Participants Continuing Buprenorphine Therapy After 6 Months of Induction
Description: After induction, clinical team will continue to follow up with patients to see if they would like to continue buprenorphine therapy during the next 6 months after induction. The date of discontinuation and the reason why will be recorded. The number of participants reported in the outcome is the number of participants that continued buprenorphine therapy 6 months after induction.
Time Frame: 6 months after induction
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Arm
Number analyzed (Participants) | 43
Participants | 38

ADVERSE EVENTS:
Time Frame: Within 72 hours of induction
Arm/Group | Buprenorphine Arm
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 1/47
Other Adverse Events (participants affected / at risk) | 9/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Arm (N=47)
Hospitalization (Nervous system disorders) | 1 (1) — Central Retinal Artery Occlusion- Thought unlikely to induction
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Arm (N=47)
Opioid Withdrawal (Psychiatric disorders) | 2 (2) — Participants with recurrent withdrawal who had their doses adjusted upward within two days.
Body Pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Participant presented with worsened pain. Participant reported pain crisis after uneventful induction.
Neck Swelling (General disorders) | 1 (1) — participant who presented with neck swelling
Tongue numbness (General disorders) | 1 (1) — participant experienced tongue numbness during induction
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Participant was admitted to the hospital for pneumonia and suspicion of delayed type hemolytic transfusion reaction related to a prior transfusion
Headache (General disorders) | 1 (1) — participant had headache during induction
Hyperglycemia (Endocrine disorders) | 1 (1) — participant with brittle type I diabetes mellitus and poor insulin adherence presenting with hyperglycemia as was typical of many prior episodes
Nausea (Gastrointestinal disorders) | 1 (1) — participant with brittle type I diabetes mellitus and poor insulin adherence presenting with nausea as was typical of many prior episodes

LIMITATIONS AND CAVEATS:
The study was not randomized nor controlled. The participant pool was limited to those patients who consented to have their data reported; and among those prospectively enrolled, to those who accepted induction. In addition, not all inductions followed the same procedure. In particular, those that were performed inpatient might have a number of biases in patient selection and capacity to detect adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT03492099/Prot_SAP_000.pdf